CLINICAL TRIAL: NCT03858218
Title: Psychometric Properties of the Chinese Version of the Pittsburgh Sleep Quality Index in Hong Kong Chinese Childhood Cancer Survivors
Brief Title: Validation of the Chinese Version of the Pittsburgh Sleep Quality Index in Hong Kong Childhood Cancer Survivors
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: UW 18-366
Record Dates: First submitted 2018-11-06; First posted 2019-02-28 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Health-Related Quality Of Life
Keywords: Psychometric properties; Sleep disturbance; Childhood cancer survivors; Quality of life,; Confirmatory factor analysis
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pediatric cancer survivors group: Childhood cancer survivors refers to those who have completed cancer treatment for at least six months, the pediatric cancer survivors must be aged 9 - 17 years, and able to communicate in Cantonese and read Chinese.This group will be required to fill in the questionnaires set.
  Interventions: Other: questionnaires set
- Healthy children group: Healthy children must be aged 9 - 17 years, and able to communicate in Cantonese and read Chinese. This group will be required to fill in the questionnaires set.
  Interventions: Other: questionnaires set

INTERVENTIONS:
Other: questionnaires set — questionnaires set: The Chinese version of the Pittsburgh Sleep Quality Index (PSQI)+The Chinese version of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC)+ The Chinese version of the Pediatric Quality of Life Inventory 4.0 Generic Core Scale (PedsQL 4.0)

SUMMARY:
Cancer is one of the major causes of death in pediatric population. In Hong Kong, childhood cancer remains a significant concern in healthcare system because of its damaging impacts on adolescent's physical and psychological functions throughout their lifespan. Particularly, adolescents surviving cancer still have to bear the health burden of numerous sequelae, even their treatment is completed for months and even years.

One of the most prevalent symptoms reported by patients surviving cancer is sleep disturbance. The causes of sleep disturbance are multifactorial. However, it can largely be attributed to disruption of circadian rhythm by prolonged use of medications and long-term hospitalization. Experiencing sleep disturbance can be devastating for survivors of cancer and precipitates inflammation and oxidative stress, which are known to be a contributing factor of neurocognitive impairment. Sleep disturbance can also lead to fatigue, which in turn limits patients' capacity in engaging in daily activities and even results in depression, severely compromising patients' quality of life in the long run. Having a reliable and valid instrument that can precisely assess the problem of sleep disturbance of cancer survivors is therefore crucial for the development and evaluation of the intervention.

The Pittsburgh Sleep Quality Index (PSQI) is the most commonly and frequently used instrument to assess sleep disturbance. Because of differences in culture and language, some concepts or items in the English version may be inappropriate for adolescents living in Hong Kong. Moreover, the psychometrics of the PSQI has only been established in adolescents undergoing active treatment for cancer, when they experienced the most severe problem. It is therefore unclear whether the PSQI can also be used to assess sleep disturbance of adolescents who have completed cancer treatment. This lack of validated instruments precludes us from understanding the severity of the problem. Also, it hinders the development of appropriate interventions that promote sleep quality. This study aims to bridge the gap in existing literature by translating the PSQI from English into Chinese, and examining the psychometrics of the translated PSQI in Hong Kong Chinese childhood cancer survivors.

DETAILED DESCRIPTION:
Cancer is one of the major causes of death in pediatric population. In Hong Kong, 46 patients aged 0 - 19 died from cancer in 2016. Childhood cancer is not common. According to Hong Kong Cancer Registry, there are approximately 190 newly diagnosed cases of childhood cancer each year. Despite this figure is not as high as that in adults, childhood cancer remains a significant concern in healthcare system because of its damaging impacts on children's physical and psychological functions throughout their lifespan. Particularly, children surviving cancer still have to pay a high price for numerous sequelae, notwithstanding their treatment is completed after months and even years.

One of the most prevalent symptoms reported by patients surviving cancer is sleep disturbance. A systematic review indicates 25 - 59 % adults reporting sleep disturbance after their treatment for cancer. A retrospective cohort study in the West also pointed out that 16.7% of childhood cancer survivors complained of disrupted sleep. The causes of sleep disturbance are multifactorial. However, it can largely be attributed to disruption of circadian rhythm by prolonged use of medications and longterm hospitalization. In fact, experiencing sleep disturbance can be devastating for survivors of cancer. Previous literature indicates that sleep disturbance precipitates inflammation and oxidative stress, which are known to be a contributing factor of neurocognitive impairment. Sleep disturbance can also lead to fatigue, which in turn limits patients' capacity in engaging in daily activities and even results in depression, severely compromising patients' quality of life in the long run. In this regard, healthcare professionals, particularly oncology nurses should bear unshrinkable responsibility to intervene this symptom with appropriate interventions, with an aim of improving the survivors' sleep quality and quality of life. Having a reliable and valid instrument that can precisely assess the problem of sleep disturbance of cancer survivors is therefore crucial for the development and evaluation of the intervention.

The Pittsburgh Sleep Quality Index (PSQI) is the most commonly used instrument to assess sleep disturbance. Although this instrument was originally developed to collect subjective information about sleep habits of psychiatric patients, it has been translated into different languages, and has been extensively applied in studies on adult cancer survivors. The results of these studies generally support this instrument to be reliable and valid in assessing sleep disturbance for this group of population. Despite the growing popularity of using this instrument in adults, no studies has so far been conducted to validate the PSQI in the pediatric population, thus limiting its usefulness for children and adolescents. In fact, a comprehensive review of the literature indicated that no validated instrument is currently available for assessing sleep disturbance of childhood cancer survivors, especially in the Hong Kong Chinese context. This lack of validated instruments precludes us from understanding the severity of the problem. Also, it hinders the development of appropriate interventions that promote sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong Chinese childhood cancer survivors who have completed cancer treatment for at least six months.
* Be aged 9 - 17 years.
* Be able to communicate in Cantonese and read Chinese.

Exclusion Criteria:

* Survivors with identified cognitive or behavioral problem(s) in their medical records

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: To assess the known-group validity, 50 pediatric cancer patients and 50 healthy children will be recruited in a pediatric oncology ward and a community center, respectively. The inclusion and exclusion for the pediatric cancer patients and healthy children will be the same as those for the childhood cancer survivors.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
The score of the Pittsburgh Sleep Quality Index (PSQI) | The outcome will be collected at the baseline.
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions which measures seven aspects of sleep: (1) subjective sleep quality, (2) sleep latency, (3) sleep duration, (4) habitual sleep efficiency, (5) sleep disturbances, (6) use of sleeping medication, and (7) daytime dysfunction. The 19 self-rated items are combined to form seven component scores, each of which has a range of 0-3 points (0 indicates no difficulty, while 3 indicates severe difficulty). The seven component scores are then summed to yield one global score, with a range of 0-21 points (0 indicating no difficulty, and 21 indicating severe difficulties in all the seven areas of sleep quality).
  The principal investigator has obtained the approval for using the Chinese version of the PSQI in this study.
The score of the Center for Epidemiologic Studies Depression Scale for Children (CES-DC) | The outcome will be collected at the baseline.
  The CES-DC is used to measure the severity of depressive symptoms in children and adolescents under 18. The respondents are invited to complete the questionnaire which consists of 20 self-report items. Each of the items is rated on a 4-point Likert scale that indicates the frequency of symptoms in the past week. A score of 0 indicates "not at all"; a score of 1 indicates "a little", a score of 2 indicates "some"; and a score of 3 indicates "a lot". Four items are reverse-scored. The sum of the 20 items is then calculated to yield a total score ranging from 0-60. A score under 15 indicates mild or no depression symptoms, while a score of 15 or higher indicates a risk for depression in children and adolescents.
  The Chinese version of the CES-DC has been released to the public.
The score of the Pediatric Quality of Life Inventory (PedsQL) 4.0 Generic Core Scales | The outcome will be collected at the baseline.
  The PedsQL is a 23-item scale that measures four dimensions of health: physical functioning, emotional functioning, social functioning, and school functioning. All items are rated on a 5-point Likert scale from 0 (Never) to 4 (Almost Always). The scoring involves a 2-step process. First, the items are reverse-scored and transformed to a 0-100 scale, i.e. 0=100, 1=75, 2=50, 3=25, 4=0. The total score is then generated by computing the mean of all item scores (i.e. the sum of all items over the number of items answered). A higher score means a better pediatric quality of life.
  The principal investigator has obtained the approval for using the Chinese version of the PedsQL in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung Wiliam Li, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ho KY, Lam KKW, Xia W, Chung JOK, Cheung AT, Ho LLK, Chiu SY, Chan GCF, Li WHC. Psychometric properties of the Chinese version of the Pittsburgh Sleep Quality Index (PSQI) among Hong Kong Chinese childhood cancer survivors. Health Qual Life Outcomes. 2021 Jul 6;19(1):176. doi: 10.1186/s12955-021-01803-y. PMID 34229705